CLINICAL TRIAL: NCT00639015
Title: Phenylephrine Versus Norepinephrine in Septic Shock: Effects on Systemic and Regional Hemodynamics. A Randomized, Controlled, Trial
Brief Title: Phenylephrine in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Morelli, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1282
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Septic Shock
Keywords: Sepsis; Septic Shock; phenylephrine; norepinephrine; catecholamine
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Phenylephrine
  Interventions: Drug: Phenylephrine
- 2 (Active Comparator): Norepinephrine
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — Titrated phenylephrine to maintain mean arterial pressure between 65-75 mmHg over a period of 12 hours from the onset of septic shock.
  Arms: 1
Drug: Norepinephrine — Titrated norepinephrine to maintain mean arterial pressure between 65-75 mmHg over a period of 12 hours from the onset of septic shock.
  Arms: 2

SUMMARY:
The present study was conducted as a prospective, randomized, controlled study to compare:

* the effects of norepinephrine and phenylephrine on systemic and regional hemodynamics in patients with catecholamine-dependent septic shock
* to test the hypothesis that norepinephrine may likewise better preserve hepatosplanchnic perfusion versus phenylephrine in patients suffering from septic shock

DETAILED DESCRIPTION:
Thirty two septic shock patients requiring vasopressor support to maintain mean arterial pressure between 65 and 75 mmHg despite adequate volume resuscitation will be enrolled in the study. Patients will be randomly allocated to be treated with either a) titrated phenylephrine, b) titrated norepinephrine (control; each n = 16), to achieve a mean arterial pressure (MAP) between 65 and 75 mmHg, if necessary. Data from right heart catheterization, thermo-dye dilution catheter, gastric tonometry as well as data from organ function, will be obtained at baseline and after 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Septic shock
* Vasopressor support to maintain mean arterial pressure (MAP) between 65 and 75 mmHg despite adequate volume resuscitation (pulmonary artery occlusion pressure = 13-18 mmHg and central venous pressure = 8-12 mmHg)

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* Present cardiac dysfunction
* Present or suspected acute mesenteric ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Systemic and regional hemodynamics | during the first 12 hours from the onset of septic shock

SECONDARY OUTCOMES:
Organ functions,adverse effects | during the first 12 hours from the onset of septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, M.D., Study Director — Departement of Anesthesiology and Intensive Care of the University of Rome "La Sapienza"
Locations (1):
- Departement of Anesthesiology and Intensive Care of the University of Rome "La Sapienza" Viale del Policlinico 155, Rome, Italy

REFERENCES:
- [Derived] Morelli A, Ertmer C, Rehberg S, Lange M, Orecchioni A, Laderchi A, Bachetoni A, D'Alessandro M, Van Aken H, Pietropaoli P, Westphal M. Phenylephrine versus norepinephrine for initial hemodynamic support of patients with septic shock: a randomized, controlled trial. Crit Care. 2008;12(6):R143. doi: 10.1186/cc7121. Epub 2008 Nov 18. PMID 19017409